CLINICAL TRIAL: NCT00392002
Title: A Cluster-Randomized Study to Examine National Characteristics and Outcome Measures of GERD Patients Utilizing the PPI Acid Suppression Symptom (PASS) Test for Response [EncomPASS].
Brief Title: Examine National Characteristics & Outcome Measures of GERD Patients Using the PPI Acid Suppression Symptom (PASS) Test for Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00096; EncomPASS
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
To characterize the burden of disease in GERD patients of prescription therapy'

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, 18 years or older, diagnosis of GERD

Exclusion Criteria:

* Peptic ulcer disease, upper gastrointestinal surgery, malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2005-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To compare the improvement in burden of overall GERD symptoms after 4 weeks of treatment with Esomeprazole verses maintenance of current therapy in subjects with persistent GERD symptoms.

SECONDARY OUTCOMES:
To examine the relationship of the severity and frequency of GERD symptoms to treatment, at national, and regional levels.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Canada Medical Director, MD, Study Director — AstraZeneca
Locations (2):
- Canada (2):
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario

REFERENCES:
- [Derived] Moayyedi P, Hunt R, Armstrong D, Lei Y, Bukoski M, White R. The impact of intensifying acid suppression on sleep disturbance related to gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2013 Apr;37(7):730-7. doi: 10.1111/apt.12254. Epub 2013 Feb 21. PMID 23432146